CLINICAL TRIAL: NCT07042412
Title: Ta'am Mustadam Intervention: Promoting Sustainable Food Choices Among Young Adults in the UAEU Community
Brief Title: Ta'am Mustadam Intervention to Promote Sustainable Food Choices
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Prof. Carine Platat, Professor, United Arab Emirates University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21R097
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Food Preferences; Health Behaviour; Choice Behavior; Feeding Behaviors; Sustainable Healthy Eating Behaviour
Keywords: Sustainable food choices; Behaviour change wheel; Intervention; Sustainable diet; Young Adults
MeSH Terms: conditions — Food Preferences; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The intervention will be conducted with a group of students affiliated with the College of Medicine and Health Sciences at the United Arab Emirates University. The intervention will last for 6 weeks, followed by a one-month post-intervention follow-up to assess lasting effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will be enrolled in the Ta'am Mustadam intervention
  Interventions: Behavioral: Ta'am Mustadam Intervention

INTERVENTIONS:
Behavioral: Ta'am Mustadam Intervention — The Ta'am Mustadam intervention will be implemented over six weeks with a four-week follow-up among students in the CMHS.
  The intervention will consist of the following elements:
  1. Education: In the mornings at 9:00 AM, educational messages will be shared via WhatsApp twice weekly (Tuesdays and Fridays), dietary tips on Wednesdays, video recipes on Saturdays, and awareness videos on Sundays. Additionally, the Planetary Health Plate will be printed on a retractable banner and placed outside the entrance of the CMHS canteen.
  2. Behavioral Practice: This component engages participants withs sustainable eating habits through biweekly challenges and hands-on meal preparation activities held on Thursdays.
  3. Environmental restructuring: Daily reminders and nudges will be delivered through WhatsApp messages, timed before participants' main meals, to promote the consumption of sustainable food choices.
  Ta'am Mustadam intervention will be evaluated using RE-AIM framework.

SUMMARY:
The goal of this pilot intervention is to learn if the Ta'am Mustadam program helps young adults make more sustainable food choices. It will also explore how the program affects their food choices, knowledge, intentions, practices, and self-reported behaviors towards sustainable food choices, as well as energy and nutrient intake.

The main questions it aims to answer are:

* Does the Ta'am Mustadam program increase intake of fruits, vegetables, and plant-based foods?
* Does it reduce red and processed meat consumption?
* Does it change participants' food choice?

The minor questions it aims to answer are:

* Does it improve participants' knowledge, intentions, practices toward sustainable eating?
* Does it change participant's energy and nutrient intake?

Participants will:

* Take part in a 6-week program, followed by a 4-week follow-up
* Receive engaging educational messages &awareness videos about sustainability
* Watch interactive video recipes
* Participate in hands-on activities
* Receive daily reminders
* Complete questionnaires before, right after, and one month after the program

Researchers will use the RE-AIM framework to assess how well the program works and whether it can be applied in real-life settings.

DETAILED DESCRIPTION:
BAACKGROUND &RATIONAL:

Suboptimal diets are a major contributor to non-communicable diseases (NCDs) and premature mortality in the United Arab Emirates (UAE). NCDs-including diabetes, cancer, chronic respiratory conditions, and cardiovascular diseases-account for 77% of all deaths and 17% of premature deaths (ages 30-70) in the country. Obesity rates have doubled since 1989, reaching 31.7% among adults by 2017, reflecting an increasing burden of diet-related chronic diseases.

At the same time, the UAE faces significant environmental pressures. Water scarcity, poor soil quality, and harsh climate conditions threaten domestic food production. Rapid population growth has intensified the demand for food and water, further straining natural resources. The UAE's dependence on food imports heightens risks to food security, dietary adequacy, and environmental sustainability.

To address these interlinked issues, the UAE has launched several policy initiatives, such as the National Food Security Strategy 2051 and the UAE National Action Plan in Nutrition, aligned with regional and international frameworks. These initiatives aim to enhance health and food system resilience while supporting environmental goals.

A key proposed solution to the interlinked challenges of diet, health, and the environment is the adoption of sustainable diets. These diets aim to promote individual health while minimizing environmental impact. The EAT-Lancet Commission introduced the "planetary health diet," a mostly plant-based model that could nourish 10 billion people by 2050 without exceeding environmental limits. Reduced meat consumption is also associated with lower risks of heart disease, cancer, and premature mortality.

The limited success of existing sustainability interventions is often due to a lack of theoretical grounding. The Behaviour Change Wheel (BCW), underpinned by the COM-B model (Capability, Opportunity, Motivation - Behaviour), provides a structured framework for designing effective interventions. It incorporates 93 behavior change techniques (BCTs) and links them with policy strategies for sustainable implementation.

To evaluate such interventions, this study applies the RE-AIM framework, which examines Reach, Effectiveness, Adoption, Implementation, and Maintenance. This model offers insights into real-world feasibility and long-term impact. Unlike purely efficacy-driven studies, RE-AIM supports practical, scalable approaches to public health challenges and contributes to implementation science aimed at bridging research and practice.

OBJECTIVES:

Primary Objectives:

* To evaluate whether the intervention promotes sustainable food choices- specifically greater consumption of fruits and vegetables, plant-based foods (e.g., legumes &nuts), and reduced intake of red and processed meats-at post-intervention and 4-week follow-up.
* To assess changes in food choice motives at post-intervention and 4-week follow-up.

Secondary Objectives:

* To examine improvements in knowledge, intentions, and practices related to sustainable diets at post-intervention and 4- week follow-up.
* To assess changes in energy and nutrient intakes at post-intervention and 4- week follow-up.
* To evaluate the intervention's real-world impact using the RE-AIM framework.

STUDY DESIGN:

This 6-week pilot intervention will use a quasi-experimental pre-post design with a 4-week follow-up, targeting 80 participants at College of Medicine and Health Sciences (CMHS). The Ta'am Mustadam intervention will be designed using BCW, will consist of three core components: 1) sending educational materials &recipes through WhatsApp group, 2) behavioral practice through activities, and 3) regular reminders and nudges delivered through WhatsApp group. The intervention focuses on increasing the consumption of fruits, vegetables, and plant-based foods (e.g., legumes &nuts), and reducing the consumption of red/processed meat intake.

ETHICAL CONSIDERATION:

Ethical approval for the study was obtained from the United Arab Emirates University Human Research Ethics (ERSC_2025_6704), and permissions were obtained from relevant university authorities. The study adheres to the Declaration of Helsinki. Participants will be informed about study procedures, data collection, and their right to withdraw at any time. Informed consent will be obtained before data collection. University email addresses will be used to match questionnaires across 3 time-points, with all data kept anonymous. Participants will receive discount vouchers at the end of the intervention

DATA COLLECTION:

Data will be collected at 3 time-points: pre-intervention (1-week before the start of intervention period), post-intervention (at intervention end) and follow-up (4-week after intervention end)

ASSESSMENT TOOLS:

* General information including participants' sociodemographic data, self- reported height and weight, and details on prior nutrition education or consultation with a dietitian.
* Food choice motives using a validated Food Choice questionnaire adapted to UAE population.
* Sustainable diet-related knowledge, intentions, practices, and self-reported behaviors will be assessed using tailored, validated tools.
* Dietary intake will be evaluated via a culturally adapted Food Frequency Questionnaire (FFQ).

ELIGIBILITY:
Inclusion Criteria:

* Undergraduates &postgraduates

Exclusion Criteria:

* Not signing the informed consent
* Reporting history of food allergies or any food intolerances (e.g., celiac disease, lactose intolerance, nut allergy, etc.)
* Reporting any medical condition that might directly affect eating patterns (e.g., Type 1 or Type 2 diabetes, cardiovascular disease, Crohn's disease, Irritable bowel syndrome)
* Under medication that affect eating patterns
* Being pregnant or breastfeeding
* Following a vegan or vegetarian diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Adoption of sustainable food choices measured by dietary intake | At pre-intervention (1-week before the start of intervention period), post-intervention (at the end of the 6-week intervention period), and follow-up (4-week after intervention end)
  Dietary intake will be assessed through a validated English version of Food Frequency Questionnaire (FFQ) tailored for the UAE population. The FFQ contains 130 culture-specific food items, divided into 12 groups. For each food item, participants could select from 9 frequency categories; "never or less than once per month", "1-3 times per month", "once per week", "2 - 4 times per week", " 5 to 6 times per week", "once per day", "2-3 times per day", "4-5 times per day", "> 6 times per day".
The extent of changes in food choice motives | At pre-intervention (1-week before the start of intervention period), post-intervention (at the end of the 6-week intervention period), and follow-up (4-week after intervention end)
  Food choice motives will be assessed using validated Food Choice Questionnaire tailored for Arabic-speaking countries That questionnaire consists of 37 items assessing nine factors: (i) health; (ii) mood; (iii) convenience; (iv) eco-ethics; (v) sensory appeal; (vi) familiarity; (vii) natural content; (viii) price; and (ix) weight control. Participants will be asked to rate the importance of each item on a four-point Likert scale with 1= "not at all important", 2= "a little important", 3= "moderately important" and 4= "very important". Mean scores for each factor will be calculated for individual respondents based on their responses.

SECONDARY OUTCOMES:
Changes in knowledge towards sustainable diets | At pre-intervention (1-week before the start of intervention period), post-intervention (at the end of the 6-week intervention period), and follow-up (4-week after intervention end)
  Knowledge about sustainable diets will be assessed through participants' agreement with five statements adapted from a validated questionnaire. The total score ranges from 0 (very little knowledge) to 10 (excellent knowledge).
Changes in intentions towards sustainable diets | At pre-intervention (1-week before the start of intervention period), post-intervention (at the end of the 6-week intervention period), and follow-up (4-week after intervention end)
  Behavioral intentions will be assessed based on participants' intent to adopt more sustainable behaviors, using an adapted questionnaire. The total score ranges from 0 to 9, with higher scores indicating a greater intention to follow a sustainable diet.
Changes in practices towards sustainable diets | At pre-intervention (1-week before the start of intervention period), post-intervention (at the end of the 6-week intervention period), and follow-up (4-week after intervention end)
  The practice will be evaluated by assessing the extent to which participants practice sustainable behaviours using an adapted questionnaire. The total score ranges from 0 to 12 (indicating a greater adherence to sustainable dietary practices).
Changes in self-reported behaviors towards sustainable diets | At pre-intervention (1-week before the start of intervention period), post-intervention (at the end of the 6-week intervention period), and follow-up (4-week after intervention end)
  Self-reported behaviors will be assessed by participants' weekly consumption of 6 food groups (e.g., "How often do you consumed fruits in a typical week") using five intake frequencies ("0 times", "1-2 times", "3-4 times", "5-6 times", "seven or more times"). This measure is adapted from previously validated questionnaire developed specifically for UAE population
Changes in baseline energy and nutrient intake | At pre-intervention (1-week before the start of intervention period), post-intervention (at the end of the 6-week intervention period), and follow-up (4-week after intervention end)
  Dietary intake will be assessed through a validated English version of Food Frequency Questionnaire (FFQ) tailored for the UAE population. The FFQ contains 130 culture-specific food items, divided into 12 groups. For each food item, participants could select from 9 frequency categories; "never or less than once per month", "1-3 times per month", "once per week", "2 - 4 times per week", " 5 to 6 times per week", "once per day", "2-3 times per day", "4-5 times per day", "> 6 times per day".

OTHER OUTCOMES:
The implementation of Ta'am Mustadam intervention at individual level | At post-intervention (at the end of the 6-week intervention period)
  The implementation of Ta'am Mustadam intervention will be assessed using an evaluation form. This questionnaire contains yes/ no questions, Likert-scale questions, and an open-ended question to collect detailed feedback from participants.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine and Health Sciences, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy reasons

REFERENCES:
- See also: Development and validation of a tool to assess knowledge, attitudes, and practices toward diet sustainability — https://www.frontiersin.org/journals/sustainable-food-systems/articles/10.3389/fsufs.2024.1432057/full
- See also: Promoting sustainable food choices through the Ta'am Mustadam pilot intervention at UAE university canteen: study protocol — https://www.frontiersin.org/journals/sustainable-food-systems/articles/10.3389/fsufs.2025.1656866/full